CLINICAL TRIAL: NCT01179854
Title: Phase 2 Double-blind,Placebo-controlled Study for Evaluation of Efficiency, Safety,Tolerance and Pharmacokinetics of Different Doses of Remegal in Additional Therapy for Patients With Refractory Partial Seizures
Brief Title: Remegal Different Doses in Patients With Refractory Partial Seizures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Valexfarm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2Р/КИ/Б; 2Р/КИ/Б (Other: Ministry of Health of Russian Federation); 2Р/КИ/Б (Other: Valexfarm)
Record Dates: First submitted 2010-07-30; First posted 2010-08-11 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Drug Safety; Normal Drug Tolerance; Self Efficacy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 500 mg (Experimental): Group of active treatment of Remegal 500 mg
  Interventions: Drug: Remegal
- Remegal 750 mg (Experimental): Group of active treatment of Remegal 750 mg
  Interventions: Drug: Remegal
- Remegal 1000 mg (Experimental): Group of active treatment of Remegal 1000 mg
  Interventions: Drug: Remegal
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Remegal

INTERVENTIONS:
Drug: Remegal — Drug/ placebo
  Other Names: Remegal (beprodone)

SUMMARY:
The purpose of this study is to determine weather different doses of Remegal are effective,safety and tolerant in Additional Therapy for Patients With Refractory Partial Seizures and pharmacokinetics definition

DETAILED DESCRIPTION:
Phase II

ELIGIBILITY:
Inclusion Criteria:

1. Subject will report to have partial onset seizures for at least the last 2 years despite prior therapy with at least 2 different consecutive AEDs.
2. Subject will report an average of at least 4 partial onset seizures per 28 days prior to entry in the Baseline phase.
3. Seizure-free period will be no longer than 21 days in the 4-week period prior to entry in the Baseline phase.
4. Subject will be on stable dosage regimen of a maximum of 3 AEDs,.
5. The dosage of concomitant AED therapy will be kept constant for at least 4 weeks prior to entry into the Baseline phase.
6. 'Subject will receive information will be given time to think about their participation and will give their written informed consent.
7. Subject will be male or female between 18 and 65 years old.
8. Subject will have a diagnosis of epilepsy with simple partial seizures and/or complex-partial seizures both with or without secondary generalization according to the ILAE (1981):

   * The results of at least one prior electroencephalogram (EEG) and magnetic resonance imaging/computerized tomography scan should be consistent with the diagnosis of partial seizures.
   * In the case of simple partial seizures, only those who motor signs will be included.

Exclusion Criteria:

1. Subject with non-epileptic events including psychogenic seizures that could be confused with seizures.
2. Subject with seizures that cannot be counted due to clustering.
3. Subject with a history of primary generalized seizures.
4. Subject with a history of status epilepticus within the 12 months period prior to trial entry.
5. Subject with concomitant treatment of felbamate or previous felbamate therapy within the last 6 months prior to trial entry.
6. Subject with concomitant treatment of vigabatrin. Subjects with previous vigabatrin therapy must have had a visual field test prior to trial entry.
7. Subject with a progressive structural lesion in the central nervous system or a progressive encephalopathy.
8. Subject who received REMEGAL in a previous trial.
9. Subject currently participating or who participated within the last two months in any trial of an investigational drug or experimental device.
10. Pregnant or nursing women and/or those of childbearing potential who are not surgically sterile, two years postmenopausal or do not practice two combined methods of contraception, unless sexually abstinent, during the duration of the trial.
11. Subject with any medical or psychiatric condition, which in the opinion of the investigator could jeopardize the subject's health or would compromise the subject's ability to participate in this trial.
12. Subject with a history of chronic alcohol or drug abuse within the previous 2 years.
13. Subject with alanine amino transferase (ALT), aspartate amino transferase (AST), alkaline phosphatase, total bilirubin, or serum creatinine level more than or equal to 2 times the upper limit of normal.
14. Subject with clinically significant abnormal vital signs.
15. Subject with a known history of severe anaphylactic reaction or serious blood dyscrasias.
16. Subject with any other clinically significant disease, surgical condition or recent chronic consumption of non-AED medications (within the preceding four weeks prior to trial entry) that might reasonably have been expected to interfere with drug absorption, distribution, metabolism or excretion.
17. Subject taking one of the following medications influencing the central nervous system within four weeks prior to trial entry: neuroleptics, monoamine oxidase (MAO) inhibitors, anxiolytics, amphetamines, sedative antihistamines, tranquilizers, hypnotics, narcotic analgesics, except for medication taken as epileptic treatment.
18. Subject with confirmed clinically significant abnormality in ECG, including prolonged QTc interval.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-09; Primary Completion 2010-11 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
safety and tolerability | Jan 2010 - Dec 2010
  The primary objective of the study is to evaluate the safety and tolerability of Remegal administered concomitantly with 1 - 3 antiepileptic drugs (AEDs) in subjects who currently have uncontrolled partial seizures with or without secondary generalization.

SECONDARY OUTCOMES:
efficacy | Jan 2010 - Dec 2010
  To assess the efficacy and its association with the Remegal dosages, and to evaluate the steady-state plasma concentrations of Remegal and concomitantly orally administered AEDs

CONTACTS AND LOCATIONS:
Overall Officials: Dorogov Nikolay, MD, PhD, Principal Investigator — MUZ"City Clinic №4"
Locations (4):
- Russia (4):
  - KGUZ "U.K. Erdman Altai Regional psychiatric hospital", Barnaul
  - Republican Dispensary, Saransk
  - GOU VPO Volgograd State medicine university of roszdrav, Volgograd
  - Sverdlovsk Regional Hospital, Yekaterinburg